CLINICAL TRIAL: NCT06199934
Title: Effectiveness of BNT162b2 Formulations Using State Vaccine Registry and Insurance Claims Data
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591065; RAVEN (Other: Alias Study Number)
Record Dates: First submitted 2023-12-18; First posted 2024-01-10 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: SARS-CoV-2; COVID-19 Vaccines
Keywords: COVID-19; XBB vaccine effectiveness
MeSH Terms: conditions — COVID-19 | interventions — Vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vaccinated: BNT162b2 recipients
  Interventions: Biological: Vaccination
- Unvaccinated: BNT162b2 eligible but did not receive

INTERVENTIONS:
Biological: Vaccination — BNT162b2 vaccination
  Groups: Vaccinated

SUMMARY:
The primary purpose of this study is to learn about how well different versions of the Pfizer-BioNTech COVID-19 vaccine (called BNT162b2) work at preventing death, severe COVID-19 that requires a trip to the hospital, and overall use of healthcare resources, such as needing to go the doctor or urgent care due to illness. Pfizer is not enrolling any participants for this study. Instead, existing data from different health data sources will be used to help answer the scientific questions Pfizer is interested in learning more about.

ELIGIBILITY:
Inclusion Criteria:

* People with at least one year of pharmacy and medical enrollment in HealthVerity prior to vaccine availability
* State of California or Louisiana resident for at least one year

Exclusion criteria:

* People currently pregnant,
* Individuals with discrepancies in sex and/or year of birth between HealthVerity claims and California/Louisiana immunization registry datasets
* A diagnosis of COVID-19 in any setting ≤ 90 days prior to start of study or receipt COVID-19 vaccine ≤ 90 days prior to start of study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were California or Louisiana residents in the HealthVerity claims database will be defined using the following hierarchical definition:
  1. Persons who have their enrollment file record indicating a patient location of California or Louisiana in HealthVerity claims enrollment file.
  2. Persons who have a patient state location other than California or Louisiana in HealthVerity claims enrollment but have one or more records in the California or Louisiana Immunization Registry. Examples include people who previously lived in Texas but moved to California and received a vaccine, or persons who crossed state lines for a vaccine and remain in their non-California state in claims data.
Sampling Method: Non-Probability Sample
Enrollment: 19853610 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Global Headquarters, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Andersen KM, McColgan MD, Mateus JS, Yu T, Zhou A, Puzniak L, Lopez SMC. BNT162b2 XBB.1.5-Adapted Single Dose Vaccine Uptake and Effectiveness in Children Aged 5-17 Years Using Linked Claims and Vaccine Registries in California and Louisiana. J Pediatr. 2025 Nov;286:114778. doi: 10.1016/j.jpeds.2025.114778. Epub 2025 Aug 14. PMID 40818804
- [Derived] Andersen KM, Allen KE, Nepal RM, Mateus JS, Yu T, Zhou A, Porter TM, Lopez SMC, Puzniak L, McLaughlin JM, McGrath LJ. Effectiveness of BNT162b2 XBB.1.5 vaccine in immunocompetent adults using tokenization in two U.S. states. Vaccine. 2025 Apr 11;52:126881. doi: 10.1016/j.vaccine.2025.126881. Epub 2025 Feb 22. PMID 39987879
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591065

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from adult and pediatric participants who were residents of California or Louisiana were collected from immunization registry linked to closed claims from HealthVerity in this retrospective study. Data was collected from HealthVerity Database from 11-Sep-2023 to 12-Mar-2024, available data was evaluated from 07-Feb-2024 to 31-Jul-2024.
Pre-assignment Details: A total of 19853610 participants were enrolled this study.
Groups:
- All Participants: Adult and pediatric participants data were collected from immunization registry linked to closed claims from HealthVerity and who were California or Louisiana residents were included.
Period: Overall Study
Arm/Group | All Participants
Started | 19853610
Completed | 19853610
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Here "Number Analyzed" signifies number of participants evaluable for this baseline characteristic.
  Years
    number analyzed (Participants) | 19702014
    (all) | 38.4 (22.03)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 10455294
  Male | 9340840
  Unknown/missing | 57476
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants COVID-19 Diagnosis
Description: Number of participants diagnosed with COVID-19 were reported in this outcome measure.
Time Frame: From date of FDA authorization/approval of BNT162b2 until end of follow-up (maximum of 6 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
Participants | 210902

2. Secondary Outcome: Number of Participants With an Outpatient Encounter
Description: Outpatient encounter was considered as an encounter with International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) code: U07.1.
Time Frame: From date of FDA authorization/approval of BNT162b2 until end of follow-up (maximum of 6 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
Participants | 130171

3. Secondary Outcome: Number of Participants With an Inpatient Encounter
Description: Inpatient encounter was considered as an encounter with ICD-10-CM code: U07.1.
Time Frame: From date of FDA authorization/approval of BNT162b2 until end of follow-up (maximum of 6 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
Participants | 11172

4. Secondary Outcome: Number of Participants With Emergency Department Encounter
Description: Number of emergency department encounter was considered as an encounter with ICD-10-CM code: U07.1.
Time Frame: From date of FDA authorization/approval of BNT162b2 until end of follow-up (maximum of 6 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
Participants | 28010

5. Secondary Outcome: Number of Participants With COVID-19 Critical Illness
Description: COVID-19 critical illness was defined as intensive care unit [ICU] admission, mechanical ventilation, or inpatient death.
Time Frame: From date of FDA authorization/approval of BNT162b2 until end of follow-up (maximum of 6 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
Participants | 3905

6. Secondary Outcome: Number of Participants With Non-COVID-19 Respiratory Infection
Description: Non-COVID-19 respiratory infection included: diagnosis of any of pneumonia, respiratory syncytial virus (RSV), rhinovirus and/or receipt of antibiotic prescription.
Time Frame: From date of FDA authorization/approval of BNT162b2 until end of follow-up (maximum of 6 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
Participants | 1869819

7. Secondary Outcome: Number of Participants With Negative Control Outcomes
Description: Negative outcomes included: accidental injury, ingrown toenail and atopic dermatitis. Number of participants with any negative control outcomes were reported in this outcome measure.
Time Frame: From date of FDA authorization/approval of BNT162b2 until end of follow-up (maximum of 6 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
Participants | 433934

8. Secondary Outcome: Total Costs of All-cause Hospitalizations From Administrative Healthcare Claims Dataset
Time Frame: From 1 month after index date (hospitalization date) until end of follow-up (Up to 4 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
US Dollars | 1008.21 (8591.93)

9. Secondary Outcome: Average Length of Stay (LOS)
Description: Average length of stay was defined as date of service end minus date of service start.
Time Frame: From 1 month after index date (hospitalization date) until end of follow-up (Up to 4 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
Days | 6.11 (7.99)

10. Secondary Outcome: Number of Participants With ICU Admission Are Included in This Outcome Measure.
Description: Percentage of participants with ICU admission within 30 Days of follow-up are included in this outcome measure.
Time Frame: From 1 month after index date (hospitalization date) until end of follow-up (Up to 4 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
Participants | 2864

11. Secondary Outcome: Number of Participants Who Received High-flow Oxygen or Mechanical Ventilation (MV)
Time Frame: From 1 month after index date (hospitalization date) until end of follow-up (Up to 4 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
Participants | 863

12. Secondary Outcome: Number of Participants With Inpatient Mortality
Time Frame: From 1 month after index date (hospitalization date) until end of follow-up (Up to 4 months)
Population: Data was not collected for this outcome measure as mortality information in the HealthVerity data was delayed several months behind real time, to protect confidentiality, and were not available at the time of analyses for the study period.
Arm/Group | All Participants
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants Who Received Antiviral Treatment
Description: Number of participants who received antiviral COVID treatment is reported.
Time Frame: From 1 month after index date (hospitalization date) until end of follow-up (Up to 4 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
Participants | 41774

14. Secondary Outcome: Mean Cost of All-cause Healthcare From Administrative Healthcare Claims Dataset
Time Frame: From 1 month after index date (hospitalization date) until end of follow-up (Up to 4 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
US Dollars | 9563.85 (134821.30)

15. Secondary Outcome: All-cause Healthcare Resource Utilization as The Total Number of Encounters, Regardless of Setting, Using Data From Administrative Healthcare Claims Dataset
Time Frame: From 1 month after index date (hospitalization date) until end of follow-up (Up to 4 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Mean (Standard Deviation); unit: Encounters
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
Encounters | 10.04 (19.85)

16. Secondary Outcome: Number of Participants With COVID-19-Related Hospitalization
Time Frame: From 1 month after index date (hospitalization date) until end of follow-up (Up to 4 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 19853610
Participants | 12129

ADVERSE EVENTS:
Time Frame: Adverse events and death were not collected; hence, time frame was not applicable
Description: In this observational retrospective study of deidentified database individual identifying information was not available. Minimum criteria for reporting an adverse event could not be met, hence SAEs and other AEs were not planned to be collected and reported.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT06199934/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT06199934/SAP_001.pdf